CLINICAL TRIAL: NCT04175119
Title: Tracking Information Flow in the Brain: A Unified and General Framework for Dynamic Communication in Brain Networks
Brief Title: Tracking Information Flow in the Brain
Acronym: BRAINDYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0854; 2019-A01604-53 (Other: ID-RCB)
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study group (Experimental): All participants signed up for experiment 1, 2, or 3 complete the same protocol (1 study arm) with an intent for intra-subject correlational analyses.
  Interventions: Device: Visual attention/perception tasks in healthy participants

INTERVENTIONS:
Device: Visual attention/perception tasks in healthy participants — The participants complete visual attention and perception tasks while fMRI, EEG, and MEG record brain signals. The tasks acquire responses with a visual saccade or button presses which are coupled to brain responses. These responses are then analyzed to identify patterns of communication between brain areas (within-subject). The flickering stimuli (experiment 1) may alter oscillations in the brain, while participants complete visual attention and perception tasks, leading to a secondary outcome measure distinct from the button presses. The procedure concerning the flickers will be the same for participants. The tACS (experiment 2) delivers input in addition to gathering output while participants complete visual attention and perception tasks. A sinusoidal current at a chosen frequency interacts with the brain's natural oscillations and alters responses. Participants will have sham sessions of tACS as well (there is no group division), The sham will be compared with the stimulation

SUMMARY:
The brain is composed of a set of areas specialized in specific computations whose outputs need to be transferred to other specialized areas for cognition to emerge. To account for context-dependent behaviors, the information must be flexibly routed through the fixed anatomy of the brain. The aim of this project is to test a general framework for this flexible communication between brain areas based on nested oscillations. The general idea is that internally-driven slow oscillations (<20Hertz) either set-up or prevent the communication between brain areas. Stimulus-driven gamma oscillations (>30Hertz), nested in the slow oscillations, can then be directed to task-relevant areas of the network. This multimodal, multi-scale approach uses magnetoencephalography using a 3-Dimensional (3D) printed individual head-cast system and transcranial stimulation in experiments manipulating visual processing, attention and memory to test core predictions of this framework. The theoretical approach and the methodological development used in this basic science study will provide the basis for future fundamental and clinical research.

ELIGIBILITY:
Inclusion Criteria:

* 20-36 years old
* Right handed
* Registered with the French healthcare system
* Motivated to participate in the study
* Normal or corrected vision
* Adequate knowledge of French to be able to follow directions and give informed consent
* Capacity to listen and follow study instructions
* Use of contraception (in sexually active women)
* BMI between 18.5 and 30
* Informed consent for participation in the study

Exclusion Criteria:

* For All Experiments:
* Persons with :

  * Sleep disorders, neurological or psychiatric illnesses or a history of such problems that could impact quality/variability of data or cooperation and retention of the subject in the study
  * Migraines or light-sensitive epilepsy
  * Regular use of medications that impact the central nervous system
  * Regular use of medications, such as opioids and antidepressants, including Selective serotonin reuptake inhibitors (SSRIs) and tricyclic antidepressants
  * Severe hearing loss
  * Skin conditions or allergies
  * Chronic pain, or any other medical conditions conducive to pain sensitivity
  * A history of stroke or recent trauma to the head
  * A pacemaker, insulin or other pump, neurostimulator, cochlear implants or other hearing aid, metal stents, prosthesis, or implants, intracerebral clips, implantable defibrillator, cerebral shunt or ventricular catheter, other foreign metal objects in the upper part of the body
* Persons unable to adhere to abstinence from the use of drugs or alcohol the day or evening before experimental sessions
* Women who are pregnant, breastfeeding, or have given birth in the last 6 months

For experiments using magnetoencephalography:

* Persons with

  * claustrophobia
  * any dental apparatus containing metal including or root canals
  * any foreign metallic object anywhere in the body
  * bolts, screws
  * orthopedic devices or implants
  * glasses (given the participant cannot use contact lenses)
  * a head size incompatible with the use of a personalized 3D head-cast or a magnetoencephalograph
* Persons having had any surgery prior to the study which puts them at risk for metal objects left in the body

For experiments using Magnetic Resonance Imaging (MRI) or Functional Magnetic Resonance Imaging (fMRI) techniques:

* Anxious, non-cooperative, or agitated persons
* Claustrophobia
* Persons having had any surgery prior to the study which puts them at risk for metal objects left in the body

For experiments using transcranial stimulation:

-Persons with frequent syncope episodes (loss of consciousness) as a result of any particular sensorial stimulations

Ages: 20 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
The composite characteristics of the brain oscillations (frequency, synchronization, and interaction between brain oscillations in and between different brain regions and networks) | up to 17 months
  The primary outcome measure is measured using fMRI bold signals (experiment 1), and brain signals obtained through electroencephalography (experiment 1, 3) and magnetoenecephalography (experiment 1, 3), depending on the sessions. The signals are then transformed during analyses and patterns in the composite characteristics are identified.

SECONDARY OUTCOMES:
The coupling of behavioral responses to stimuli with physiological responses in the brain. | up to 17 months
  Throughout the sessions of neuroimaging. There are 5, 1 or 2, and 1 sessions of neuroimaging for experiment 1, 2, and 3 respectively. The 5 sessions of experiment 1 are over a period of 1 to 17 months. Each session lasts approximately 3 hours including setup.The sessions take place at between 7 and 198 days after inclusion. The time between the sessions is variable.
Coupling of brain oscillation characteristics in responses to the "flickering" effect | up to 17 months
  There are 5 sessions of neuroimaging for experiment 1. The 5 sessions of experiment 1 are over a period of 1 to 17 months. Each session lasts approximately hours including setup. This outcome measure will be recorded during these 5 interspaced sessions, at between 7 and 198 days after inclusion. The time between the sessions is variable.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Bonnefond, PhD, Principal Investigator — INSERM Rhône Alpes
Locations (1):
- Centre de Recherche en Neuroscience de Lyon INSERM, Bron, France